CLINICAL TRIAL: NCT06596252
Title: Double-blind, Randomized, Non-inferiority Phase III Trial on the Efficacy and Tolerability of 2 mg Once Daily vs. 1 mg Twice Daily Budesonide Orodispersible Tablets in Adults With Eosinophilic Esophagitis
Brief Title: Once Daily Versus Twice Daily Budesonide Orodispersible Tablets for Induction of Remission in EoE
Acronym: EOS-4
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BUL-8/EEA; 2024-515229-26-00 (EU CTIS Number); 2020-001314-37 (EudraCT Number)
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Eosinophilic Esophagitis
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Budesonide 2 mg orodispersible tablet once daily
  Interventions: Drug: Budesonide
- Arm B (Active Comparator): Budesonide 1 mg orodispersible tablet twice daily
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — Twice daily intake of the tablet 30 min after a meal

SUMMARY:
The purpose of this study is to prove the non-inferiority of a 6-weeks treatment with 1 mg budesonide orodispersible tablets BID versus 2 mg budesonide orodispesible tabletss for the induction of clinico-pathological remission in adult patients with active eosinophilic esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent,
* Male or female patients, 18 to 75 years of age,
* Confirmed clinico-pathological diagnosis of eosinophilic esophagitis (EoE) according to established diagnostic criteria
* Active symptomatic and histological EoE
* Negative pregnancy test in females of childbearing potential at baseline visit.

Exclusion Criteria:

* Clinical and endoscopic signs of gastroesophageal reflux disease (GERD),
* Achalasia, scleroderma esophagus, or systemic sclerosis,
* Other clinically evident causes than EoE for esophageal eosinophilia,
* Any concomitant esophageal disease and relevant gastro-intestinal disease (celiac disease, inflammatory bowel disease, oropharyngeal or esophageal bacterial, viral, or fungal infection [candida esophagitis]),
* Any relevant systemic disease (e.g., AIDS, active tuberculosis, hepatitis B or C),
* If careful medical monitoring is not ensured: cardiovascular disease, diabetes mellitus, osteoporosis, active peptic ulcer disease, glaucoma, cataract, or infection,
* Liver cirrhosis or portal hypertension,
* History of cancer in the last five years,
* History of esophageal surgery at any time or of esophageal dilation procedures within the last 4 weeks prior to screening visit, or need for an immediate endoscopic intervention due to a stricture
* Upper gastrointestinal bleeding within 8 weeks prior to baseline visit,
* Existing or intended pregnancy or breast-feeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in histological remission | 6 weeks
  Histological assessment of biopsies taken at end of treatment visit

SECONDARY OUTCOMES:
Proportion of patients in clinical remission | 6 weeks
  Assessment of clinical scores assessed with questionnaires at the end of treatment visit

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo J Lucendo, MD, PhD, Study Director — Department of Gastroenterology, Hospital General de Tomelloso, Spain
Locations (14):
- United States (13):
  - Dr. Falk Investigational Site, La Jolla, California
  - Dr. Falk Investigational Site, Lomita, California
  - Dr. Falk Investigational Site, Boise, Idaho
  - Dr. Falk Investigational Site, Houma, Louisiana
  - Dr. Falk Investigational Site, Marrero, Louisiana
  - Dr. Falk Investigational Site, Boston, Massachusetts
  - Dr. Falk Investigational Site, Rochester, Minnesota
  - Dr. Falk Investigational Site, Freehold, New Jersey
  - Dr. Falk Investigational Site, Jackson, New Jersey
  - Dr. Falk Investigational Site, Chapel Hill, North Carolina
  - Dr. Falk Investigational Site, Cleveland, Ohio
  - Dr. Falk Investigational Site, Harlingen, Texas
  - Dr. Falk Investigational Site, Salt Lake City, Utah
- Department of Gastroenterology, Hospital General de Tomelloso, Tomelloso, Spain

IPD SHARING:
Plan to Share IPD: Yes
It is not yet decided which data will be made available. Neither a time frame can be indicated yet.
Time Frame: It is not yet decided which data will be made available. Neither a time frame can be indicated yet.
Access Criteria: Contact to Dr. Falk, issue of confidentiality agreement for any information not publicly available.